CLINICAL TRIAL: NCT00244907
Title: Metabolism and Bone Health
Brief Title: Isoflavones for Promoting Calcium Absorption and Preventing Bone Loss in Post Menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Office of Dietary Supplements (ODS) (NIH)
Responsible Party: Principal Investigator, Berdine Martin, Research Scientist, Nutrition Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: P50AT000477-06 (NIH); P50AT000477-06 (NIH)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Bone Resorption; Phytoestrogens; Calcium; Genistein; Equol
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Bone Resorption | interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Genistein vs. Risedronate (Active Comparator): Healthy post menopausal women who have been dosed with Ca41. Intervention, 100 mg Gensitein from soy protein isolate for 50 days. After a 50 day washout risedronate (Actonel- 5mg per day) for 50 days
  Interventions: Dietary Supplement: Genistein vs Risedronate
- Genistein dose and source (Active Comparator): Healthy post menopausal women will consume 5 products containing varying quantities of genistein from different sources for 50 days each in a randomized order. Each intervention period is separated by a 50 day washout period. Intervention: A) 50 mg genistein from soy protein isolate, B) 100 mg genistein from soy protein isolate, C)50 mg genistein from Novasoy, D) 100 mg genistein from Novasoy, E) 100 ng genistein from 50% Novasoy and 50% soy protein isolate
  Interventions: Dietary Supplement: Genistein vs Risedronate

INTERVENTIONS:
Dietary Supplement: Genistein vs Risedronate — Gensitein (100 gm) from soy protein isolate Risedronate (5 mg)
  Other Names: Actonel

SUMMARY:
Estrogen is a hormone that helps prevent calcium loss and bone breakdown. During menopause, estrogen levels decrease. Insufficient amounts of estrogen may lead to bone loss and possibly osteoporosis. Isoflavones are natural compounds found in soy plants that may help provide protection against bone loss. This study will evaluate the effect of soy isoflavones on calcium absorption and bone loss in post menopausal women.

DETAILED DESCRIPTION:
Estrogen is a hormone that activates bone-forming cells and prevents calcium loss and bone breakdown. During menopause, estrogen levels decrease. Insufficient amounts of estrogen may accelerate bone breakdown and inhibit the body's ability to create new bone, thereby leading to bone loss and possibly osteoporosis. Various treatments have been developed to decrease bone loss in post-menopausal women. Actonel, for example, is an FDA-approved drug used to help prevent bone loss.

Phytoestrogens are plant compounds with a structure similar to estrogen. They have also been shown to help reduce the negative effects of menopause. Isoflavones are a particular type of phytoestrogens that are found in soy plants and may act like estrogen in providing possible protection against bone loss. This study will compare the effects of isoflavones (including genistein, a type of isoflavone) versus Actonel on calcium absorption and bone loss in post-menopausal women.

Participants in this double-blind cross-over study will first complete a screening process, which will include answering questions about their health habits, medical history, physical activity, and food patterns. They will then eat one soy bar daily for 3 days. On Day 4, a urine sample will be taken to assess their ability to metabolize phytoestrogen from soybeans. Participants will be randomly assigned to a specific treatment order. Participants will receive 1-4 unique soy isoflavones, followed by Actonel. Treatment phases will be separated by a 50-day washout period. All participants will also take calcium and vitamin D supplements throughout the study. Assessments will include bone density measurements, calcium absorption tests, and blood and urine tests. The study will last approximately 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* At least 4 years post-menopausal

Exclusion Criteria:

* Not currently taking estrogen replacement therapy or undergoing any treatment for osteoporosis
* Diagnosis of breast cancer
* Results of mammogram suggesting breast cancer

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Urinary markers of bone resorption; measured at the end of each treatment phase | Every 50 days

SECONDARY OUTCOMES:
Serum markers of bone resorption and calcium absorption; measured at the end of each treatment phase | Every 50 days

CONTACTS AND LOCATIONS:
Overall Officials: Connie M. Weaver, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Background] Spence LA, Lipscomb ER, Cadogan J, Martin B, Wastney ME, Peacock M, Weaver CM. The effect of soy protein and soy isoflavones on calcium metabolism in postmenopausal women: a randomized crossover study. Am J Clin Nutr. 2005 Apr;81(4):916-22. doi: 10.1093/ajcn/81.4.916. PMID 15817872
- [Background] Jackson GS, Weaver C, Elmore D. Use of accelerator mass spectrometry for studies in nutrition. Nutr Res Rev. 2001 Dec;14(2):317-34. doi: 10.1079/NRR200129. PMID 19087429
- [Derived] Pawlowski JW, Martin BR, McCabe GP, McCabe L, Jackson GS, Peacock M, Barnes S, Weaver CM. Impact of equol-producing capacity and soy-isoflavone profiles of supplements on bone calcium retention in postmenopausal women: a randomized crossover trial. Am J Clin Nutr. 2015 Sep;102(3):695-703. doi: 10.3945/ajcn.114.093906. Epub 2015 Aug 5. PMID 26245807
- [Derived] Nakatsu CH, Armstrong A, Clavijo AP, Martin BR, Barnes S, Weaver CM. Fecal bacterial community changes associated with isoflavone metabolites in postmenopausal women after soy bar consumption. PLoS One. 2014 Oct 1;9(10):e108924. doi: 10.1371/journal.pone.0108924. eCollection 2014. PMID 25271941